CLINICAL TRIAL: NCT04116918
Title: Efficacy and Safety of the Combination of Anlotinib and JS001 in EGFR-TKI Resistant T790M-Negative NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Baodong Qin (Other)
Responsible Party: Sponsor-Investigator, Baodong Qin, Clinical Resident, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Other Study IDs: AJERTNN
Record Dates: First submitted 2019-07-16; First posted 2019-10-07 (Actual); Last update posted 2019-10-07 (Actual); Status verified 2019-10

CONDITIONS: NSCLC Stage IV; EGFR T790M-negative; Anlotinib; JS001
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is designed to evaluate the efficacy and safety of the combination of Anlotinb and JS001 in EGFR-TKI resistant T790M-negative NSCLC patients.

DETAILED DESCRIPTION:
All EGFR mutation NSCLC patients with EGFR-TKIs eventually develop acquired resistance and in 40%-50% of these the resistance mechanism is based on the EGFR T790M mutation who could receive Osimertinib. Several alternative mechanisms of escape from EGFR-TKIs have been detected in NSCLC patients without the T790M, such as Met application, BRAF mutation, PIK3CA mutation, etc, who could receive the combination of EGFR-TKI with comparable target drug. Given the lack of targeted therapy for the majority of T790M-negative patients, platinum-doublet chemotherapy remains the standard of care with low effectiveness. In the present study, we aimed to evaluate the efficacy and safety of the combination of Anlotinb and JS001 in EGFR-TKI resistant T790M-negative NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients >=18 years of age
* Inoperable locally advanced, recurrent, and/or metastatic NSCLC patients with EGFR sensitive mutation
* EGFR-TKI resistent
* EGFR T790M negative
* Expected survival ≥ 3 month;
* ECOG / PS score: 0-2;
* the main organ function to meet the following criteria: HB ≥ 90g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L,BIL <1.5 times the upper limit of normal (ULN); Liver ALT and AST <2.5 × ULN and if liver metastases, ALT and AST <5 × ULN; Serum Cr ≤ 1 × ULN, endogenous creatinine clearance ≥50ml/min

Exclusion Criteria:

* EGFR-T790M positive
* with druggable gene alteration;
* Patient can not comply with research program requirements or follow-up;

Ages: 18 Months to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: EGFR-TKI Resistant T790M-Negative NSCLC
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Evaluation of tumor burden based on RECIST criteria until first documented progress through study completion, an average of 2 months
  Time from treatment beginning until disease progression
Objective Response Rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 2 months
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission.

SECONDARY OUTCOMES:
Overall Survival | From date of treatment beginning until the date of death from any cause, through study completion, an average of 1 months
  Time from treatment beginning until death from any cause
Adverse Effect | Through study completion, an average of 1 months
  Incidence of Treatment-related adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, China